CLINICAL TRIAL: NCT03838653
Title: Influence of Tracheal-bronchial Anatomy Changes on Multi-detector Computed Tomography Scan of the Chest Upon Placement of Left-Sided Double Lumen Endotracheal Tube
Status: Completed | Type: Observational
Sponsor: Javier H Campos (Other)
Responsible Party: Sponsor-Investigator, Javier H Campos, Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 201207717
Record Dates: First submitted 2019-02-05; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Intubation, Intratracheal; Multidetector Computed Tomography
Keywords: Double-lumen endotracheal tube; Multidetector Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Left main bronchus (LMB) intubation: Thoracic surgery patient is intubated with left side double lumen tube (L-DLT) and a fiberoptic bronchoscope is used to verify optimal positioning. The patient is designated as this group when the endobronchial lumen is observed to be in the left main bronchus (correct placement).
- Right main bronchus (RMB) intubation: Thoracic surgery patient is intubated with left side double lumen tube (L-DLT) and a fiberoptic bronchoscope is used to verify optimal positioning. The patient is designated as this group when the endobronchial lumen is observed to be in the right main bronchus (incorrect placement).

SUMMARY:
One-lung ventilation (OLV) is used for thoracic surgical procedures to facilitate surgical exposure. Lung isolation is performed using a double-lumen endotracheal tube (DLT) and optimal position is achieved with the use of fiberoptic bronchoscopy. The most common technique used to place a left-sided DLT is the blind method technique, which consists of direct laryngoscopy and rotation of the DLT into the trachea with the aim to intubate the entrance of the left main bronchus. The DLT will be rotated counterclockwise blindly after the tip of the DLT passes the vocal cords under direct laryngoscopy. However, in some occasions, the tip of the DLT migrates into the right bronchus because the alignment between the trachea and right bronchus is more vertical. The identification of the misplacement can be challenging, which could lead to the failure of lung isolation. In order to avoid the unsuccessful lung isolation, Investigators are interested in identifying the factors that potentially influence the incorrect tube DLT placement diverting into the opposite bronchus.

DETAILED DESCRIPTION:
Recently, multi-detector 3-dimensional computed tomography (MDCT) scan of the chest is becoming a routine study for patients requiring thoracic surgical procedures. On the day of thoracic surgery, the participant will be intubated with a left-sided DLT and investigators will confirm the correct insertion of the left-sided DLT at first pass under direct laryngoscopy. This information will be recorded and saved. After the study is completed, investigators will review the MDCT of the chest to review any abnormal findings and correlate it with the success of the insertion of the left-sided DLT into the left bronchus. Investigators will conduct a pilot study to determine the most influential anatomical change that leads to the DLT misplacement at the first pass based upon the changes of the tracheal-bronchial anatomy on MDCT.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Adult patient undergoing scheduled thoracic surgery which requires left side double lumen tube placement

Exclusion Criteria:

* More than 90 years of age
* Patients with emergency surgery
* Prisoners
* Patients who cannot provide their own consent
* Patient refusal
* Non-English speaking patients

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient undergoing scheduled thoracic surgery at University of Iowa Hospital
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2013-06-19 (Actual); Study Completion 2013-06-19 (Actual)

PRIMARY OUTCOMES:
Measure tracheal length (mm) derived from MDCT images | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. Tracheal length as seen on MDCT images will be measured (millimeters) and compared between the two groups.
Measure LMB diameter (mm) derived from MDCT images | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. The LMB as seen on MDCT images will be measured (millimeters) and compared between the two groups.
Measure RMB diameter (mm) derived from MDCT images | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. The RMB as seen on MDCT images will be measured (millimeters) and compared between the two groups.
Measure the tracheal LMB curvature (TLMBC) derived from MDCT images | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. The TLMBC as seen on MDCT images will be measured and compared between the two groups. TLMBC is measured at the Trachea LMB branch point. The center lines of the airway segments (trachea and LMB) close to the branch point are displayed. A circumscribed circle goes through three adjacent airway points centered at the branch point is produced and the curvature is calculated by the reciprocal of the circle radius. The curvature of a straight line is zero. A larger curvature indicates a sharper turning angle.
Measure the tracheal RMB curvature (TRMBC) derived from MDCT images | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. The TRMBC as seen on MDCT images will be measured and compared between the two groups. TRMBC is measured at the Trachea LMB branch point. The center lines of the airway segments (trachea and RMB) close to the branch point are displayed. A circumscribed circle goes through three adjacent airway points centered at the branch point is produced and the curvature is calculated by the reciprocal of the circle radius. The curvature of a straight line is zero. A larger curvature indicates a sharper turning angle.

SECONDARY OUTCOMES:
Calculate the TLMBC/TRMBC (TLMB/TRMB) Curvature Ratio | Within 1 month
  Participants are divided into two groups based upon the first pass location of the L-DLT; LMB (left main bronchus) intubation group and RMB (right main bronchus) intubation group. A ratio of the TLMBC and TRMBC values reported above will be calculated and compared between the two groups.
Incidence of the DLT misplacement (RMB intubation) at the fast pass | Within 10 minutes
  The number of times DLT misplacement (RMB intubation) at the first pass will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Javier H Campos, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data (IPD) collected during the trial, after de-identification will be shared with researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal. IPD will be available for sharing immediately after publication and ending 5 years following article publication.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be available for sharing immediately after publication and ending 5 years following article publication.
Access Criteria: Individual participant data will be accessible to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal